CLINICAL TRIAL: NCT04541979
Title: Aerosoliserat DNase for Treatment of Respiratory Failure in Severe COVID-19 - a Phase 2, Single-blinded, Randomized Study
Brief Title: Aerosoliserat DNase for Treatment of Respiratory Failure in Severe COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Adam Linder, senior concultant, associate professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NETSC-19
Record Dates: First submitted 2020-06-05; First posted 2020-09-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerosolized DNase I (Active Comparator)
  Interventions: Drug: aerosolized DNase
- NaCl (Placebo Comparator)
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: aerosolized DNase — DNase
  Arms: Aerosolized DNase I
Drug: NaCl — NaCl 0.9%, isotonic saline
  Arms: NaCl

SUMMARY:
Recent observations have suggested a role of neutrophil extracellular traps (NETs) in the pathophysiology of severe COVID-19. The aim of the study is to assess efficacy and safety of aerosolized DNase I to remove NETs and decrease respiratory distress in patients with COVID-19.

DETAILED DESCRIPTION:
Study objectives: Primary objective: To compare the treatment effect of aerosolized DNase I to that of placebo (NaCl, 0.9%) on time to cessation of oxygen therapy or discharge from hospital in hospitalized patients with COVID-19 and respiratory dysfunction.

Secondary objectives: To compare the treatment effect of aerosolized DNase I to that of placebo (NaCl, 0.9%) on 28-day mortality, days alive and without ventilator treatment, days alive and without high flow nasal oxygen treatment (Optiflow), length of stay in the ICU, days alive and outside hospital, relapse of hypoxia, days alive and without need for supplemental oxygen, adverse reactions.

Exploratory objectives: To compare the treatment effect of aerosolized DNase I to that of placebo (NaCl, 9%) on quantification of NETs in respiratory secretions and on the incidence of clinical thromboembolic events.

Study design: Phase 2 open-label randomized controlled multicentre trial. The study period is 28 days from randomization. A long term follow-up on mortality and readmission will also be collected via patient medical records/registries at day 90, day 180, and day 360 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Admitted to hospital ward or ICU
* A positive PCR test for SARS-CoV-2 from throat swab or nasopharynx
* An oxygen saturation ≤90% after maximum 15 minutes without supplemental oxygen
* Signed informed consent

Exclusion Criteria:

* Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation
* Known or suspected allergy against Pulmozyme
* Chronic obstructive pulmonary disease stage III-IV or another comparable chronic respiratory disease
* Participation in a clinical study with an investigational product during the last 30 days
* Previous participation in this study
* Pregnancy. Women of childbearing potential must agree to use contraceptives for the duration of the study period
* Any condition that, in the opinion of the Investigator, would place the patient at increased risk or preclude the patient's compliance with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Time to cessation of oxygen therapy DNase I to that of placebo (NaCl, 0.9%) on time to cessation of oxygen therapy hospitalized patients with COVID-19 and respiratory dysfunction. | 28 days
  Number of Days to cessation of oxygen therapy after start of treatment

SECONDARY OUTCOMES:
28-day mortality | 28 days
  Number of diseased patients up to 28 Days after start of treatment
Number of Days alive and without ventilator treatment | 28 days
  Number of Days alive and without ventilator treatment up to 28 Days after start of treatment
Number of Days alive and without high flow nasal oxygen treatment (Optiflow) | 28 days
  Number of Days alive and without high flow nasal oxygen treatment (Optiflow) up to 28 Days after start of treatment
Number of Days alive and free of stay in the ICU | 28 days
  Number of Days alive and free of stay in the ICU up to 28 Days after start of treatment
Number of Days alive and outside hospital | 28 days
  Number of Days alive and outside hospital up to 28 Days after start of treatment
Number of Days alive and free of a new episode and with oxygen saturation ≤93% after primary endpoint has been met | 28 days
  Number of Days alive and free of a new episode and with oxygen saturation ≤93% after primary endpoint has been met up to 28 Days after start of treatment
Number of Days alive and without need of supplemental oxygen | 28 days
  Number of Days alive and without need of supplemental oxygen up to 28 Days after start of treatment
Number of patients with adverse reactions | 28 days
  Number of patients with adverse reactions reported up to 28 Days after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adam Linder, MD, Principal Investigator — Region Skåne
Locations (1):
- Lund ED, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
nn